CLINICAL TRIAL: NCT04280081
Title: A Phase 2 Study of Oral Selpercatinib (LOXO-292) in Patients With Advanced Solid Tumors, Including Rearranged in Transfection (RET) Fusion-Positive Solid Tumors, Medullary Thyroid Cancer and Other Tumors With RET Activation
Brief Title: A Study of Selpercatinib (LY3527723) in Participants With Advanced Solid Tumors Including RET Fusion-positive Solid Tumors, Medullary Thyroid Cancer and Other Tumors With RET Activation
Acronym: LIBRETTO-321
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17492; J2G-GH-JZJK (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Medullary Thyroid Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Targeted Therapy; Medullary Thyroid Carcinoma; Thyroid Cancer; RET Alteration; MTC
MeSH Terms: conditions — Carcinoma, Medullary; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Selpercatinib (Experimental): Selpercatinib 160 milligrams (mg) administered orally twice daily (BID).
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292

SUMMARY:
The reason for this study is to see if the study drug selpercatinib is safe and effective in participants in China with rearranged during transfection (RET) fusion-positive solid tumors, medullary thyroid cancer (MTC) and other tumors with RET activation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a locally advanced or metastatic solid tumor.
* Evidence of a RET gene alteration in tumor and/or blood.
* Measurable or non-measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2, with no sudden deterioration 2 weeks prior to the first dose of study treatment.
* Archived tumor tissue sample available for cohort 1 and 2.
* Cohorts 1 and 2: failed or intolerant to standard of care.
* Cohorts 1-2: enrollment will be restricted to participants with evidence of a RET gene alteration in tumor (i.e., not just blood). However, a positive germline DNA test for a RET gene mutation as defined in the protocol is acceptable in the absence of tumor tissue testing for participants with MTC.
* Cohorts 1-2: at least one measurable lesion as defined by RECIST v1.1 and not previously irradiated (unless progressive disease for the irradiated lesion[s] has been radiographically documented).

Exclusion Criteria:

* Cohorts 1-2, an additional validated oncogenic driver that could cause resistance to selpercatinib treatment if known.
* Prior treatment with a selective RET inhibitor(s) (including investigational selective RET inhibitor(s), such as BLU-667, RXDX-105, etc).
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Any unresolved toxicities from prior therapy greater than common terminology criteria for adverse events (CTCAE) Grade 1 except where otherwise noted in this eligibility criteria at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum therapy-related neuropathy.
* Symptomatic primary central nervous system (CNS) tumor, symptomatic CNS metastasis, leptomeningeal carcinomatosis, or untreated spinal cord compression.
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of selpercatinib or prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 milliseconds.
* History of Human Immunodeficiency Virus (known HIV 1/2 antibodies positive); participants with unknown HIV status do not need to be tested.
* History of active hepatitis B (known positive hepatitis B surface antigen [HbsAg] and quantitative hepatitis B DNA greater than the upper limit of detection of the assay) or C (known positive hepatitis C antibody and quantitative hepatitis C RNA greater than the upper limit of detection of the assay); participants with unknown hepatitis B/hepatitis C status do not need to be tested.
* Active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing intercurrent illness, such as hypertension or diabetes, despite optimal treatment. Screening for chronic conditions is not required.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.
* Uncontrolled symptomatic hyperthyroidism or hypothyroidism
* Uncontrolled symptomatic hypercalcemia or hypocalcemia.
* Concurrent use of drugs known to prolong QTc.
* Pregnancy or lactation. Breast-feeding should be interrupted when selpercatinib is started; breast-feeding can be resumed 3 months after discontinuation of selpercatinib.
* Active second malignancy other than minor treatment of indolent cancers with prior sponsor approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2027-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM, Study Director — Eli Lilly and Company
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai/China
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Lu S, Cheng Y, Huang D, Sun Y, Wu L, Zhou C, Zhou J, Guo Y, Shao J, Zhang W. Selpercatinib in Chinese patients with RET-fusion-positive non-small-cell lung cancer: updated efficacy and safety analysis from the LIBRETTO-321 phase II trial. Ther Adv Med Oncol. 2025 Jan 1;17:17588359241307199. doi: 10.1177/17588359241307199. eCollection 2025. PMID 39759832
- [Derived] Lu S, Zheng X, Sun Y, Huang D, Wu L, Ji Q, Zhou C, Zhou J, Guo Y, Ge M, Ding D, Shao J, Zhang W, Gao M, Cheng Y. Patient-reported outcomes following selpercatinib treatment in Chinese patients with advanced RET fusion-positive non-small-cell lung cancer and thyroid cancer, and RET-mutant medullary thyroid cancer in the phase II LIBRETTO-321 trial. Ther Adv Med Oncol. 2023 Aug 25;15:17588359231189429. doi: 10.1177/17588359231189429. eCollection 2023. PMID 37655205
- [Derived] Cheng Y, Huang D, Zhou J, Zhou C, Sun Y, Wu L, Guo Y, Jingxin S, Zhang W, Lu S. Intracranial Activity of Selpercatinib in Chinese Patients With Advanced RET Fusion-Positive Non-Small-Cell Lung Cancer in the Phase II LIBRETTO-321 Trial. JCO Precis Oncol. 2023 Jun;7:e2200708. doi: 10.1200/PO.22.00708. PMID 37315261
- [Derived] Zheng X, Ji Q, Sun Y, Ge M, Zhang B, Cheng Y, Lei S, Shi F, Guo Y, Li L, Chen L, Shao J, Zhang W, Gao M. Efficacy and safety of selpercatinib in Chinese patients with advanced RET-altered thyroid cancers: results from the phase II LIBRETTO-321 study. Ther Adv Med Oncol. 2022 Aug 29;14:17588359221119318. doi: 10.1177/17588359221119318. eCollection 2022. PMID 36062046
- [Derived] Lu S, Cheng Y, Huang D, Sun Y, Wu L, Zhou C, Guo Y, Shao J, Zhang W, Zhou J. Efficacy and safety of selpercatinib in Chinese patients with advanced RET fusion-positive non-small-cell lung cancer: a phase II clinical trial (LIBRETTO-321). Ther Adv Med Oncol. 2022 Jul 28;14:17588359221105020. doi: 10.1177/17588359221105020. eCollection 2022. PMID 35923928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this study was based on tumor type.
Pre-assignment Details: Primary analysis set (PAS) is defined as rearranged transfection (RET) fusion positive non-small cell lung cancer (NSCLC) and thyroid cancer (TC) and RET mutant medullary thyroid cancer (MTC). Enrolled population is defined as all eligible participants.
Groups:
- Selpercatinib: 160 milligram (mg) Selpercatinib administered orally twice daily (BID).
Period: Overall Study
Arm/Group | Selpercatinib
Started | 77
Enrolled: All NSCLC | 47
Enrolled: All TC | 1
Enrolled: All MTC | 29
PAS: RET Fusion Positive NSCLC | 26
PAS: RET Fusion Positive TC | 1
PAS: Advance RET-mutant MTC | 26
Completed | 65
Not Completed | 12
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Progressive Disease | 6

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Selpercatinib: 160 mg Selpercatinib administered orally BID.
Arm/Group | Selpercatinib
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.60 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 77
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 77

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis Set: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR) as Assessed by Independent Review Committee (IRC)
Description: ORR is the summary measure of best overall response (BOR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. BOR is defined as the best response designation for each participant that is recorded between the date of the first dose of selpercatinib and the date of documented disease progression per RECIST 1.1 or the date of subsequent therapy, whichever occurs first, and subsequently confirmed. BOR will be categorized as complete response (CR), partial response (PR). CR is defined as Disappearance of all target lesions. Any pathologic nodes (whether target or non-target lesions) must have a reduction in short axis diameter (SAD) to less than 10 mm. PR At least 30% decrease in the sum of the diameters (SOD) (LD for non-nodal lesions and SAD for nodal lesions) of target lesions, taking as reference the baseline sum LD.
Time Frame: Date of First Dose to Disease Progression or Death (up to 12 Months)
Population: All treated participants who have confirmed RET fusion positive solid tumor NSCLC,TC, or RET mutant MTC by central lab, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RET Fusion Positive Non-small Cell Lung Cancer (NSCLC) Cohort 1; RET Fusion Positive Thyroid Cancer (TC) Cohort 1; RET Mutant Medullary Thyroid Cancer (MTC) Cohort 2: 160 mg Selpercatinib administered orally BID.
Arm/Group | RET Fusion Positive Non-small Cell Lung Cancer (NSCLC) Cohort 1 | RET Fusion Positive Thyroid Cancer (TC) Cohort 1 | RET Mutant Medullary Thyroid Cancer (MTC) Cohort 2
Number analyzed (Participants) | 26 | 1 | 26
percentage of participants
  Complete Response | 3.8 [0.1 to 19.6] | 0 [0.0 to 97.5] | 7.7 [0.9 to 25.1]
  Partial Response | 65.4 [44.3 to 82.8] | 100.0 [2.5 to 100.0] | 50.0 [29.9 to 70.1]
  Overall Response (CR/PR) | 69.2 [48.2 to 85.7] | 100.0 [2.5 to 100.0] | 57.7 [36.9 to 76.6]

2. Primary Outcome: Enrolled Population: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR) as Assessed by IRC
Description: as for outcome 1
Time Frame: Date of First Dose to Disease Progression or Death (Up to 12 months)
Population: All eligible participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Non-small Cell Lung Cancer (All NSCLC); Thyroid Cancer (All TC); Medullary Thyroid Cancer (All MTC): 160 mg Selpercatinib administered orally BID.
Arm/Group | Non-small Cell Lung Cancer (All NSCLC) | Thyroid Cancer (All TC) | Medullary Thyroid Cancer (All MTC)
Number analyzed (Participants) | 47 | 1 | 29
percentage of participants
  Complete Response | 6.4 [1.3 to 17.5] | 0 [0.0 to 97.5] | 10.3 [2.2 to 27.4]
  Partial Response | 59.6 [44.3 to 73.6] | 100.0 [2.5 to 100.0] | 48.3 [29.4 to 67.5]
  Overall Response (CR/PR) | 66.0 [50.7 to 79.1] | 100.0 [2.5 to 100.0] | 58.6 [38.9 to 76.5]

3. Secondary Outcome: Enrolled Population: Duration of Response (DoR) as Assessed by IRC
Description: DOR is defined as the number of months from the start date of PR or CR (whichever response is recorded first), and subsequently confirmed, to the date of disease progression or death, whichever occurs earlier.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Up to 11 Months)
Population: All eligible participants with confirmed response. Number of participants censored: All NSCLC = 30, All TC = 1, and All MTC = 16.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All NSCLC; All TC; All MTC: 160 mg Selpercatinib administered orally BID.
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 31 | 1 | 17
months | NA [NA to NA] — Median not evaluable due to number of participants censored. | NA [NA to NA] — Median not evaluable due to number of participants censored. | NA [NA to NA] — Median not evaluable due to number of participants censored.

4. Secondary Outcome: Enrolled Population: Time to Response (TTR) as Assessed by IRC
Description: TTR is defined as the number of months elapsed between the date of the first dose of selpercatinib and the first documentation of objective response (CR or PR, whichever occurs earlier) that is subsequently confirmed.
Time Frame: Date of First Dose to First Occurrence of Confirmed Tumor Response (Up to 6 months)
Population: All eligible participants with confirmed response.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 31 | 1 | 17
months | 1.84 [1.74 to 1.87] | 1.74 [1.74 to 1.74] | 1.84 [1.81 to 3.71]

5. Secondary Outcome: Enrolled Population: Time to Best Response (TTBR) as Assessed by IRC
Description: as for outcome 4
Time Frame: Date of First Dose to First Occurrence of PR (If Subject's Best Overall Response [BOR] is PR) or CR (If Subject's BOR is CR) (Up to 8 months)
Population: All eligible patients with confirmed response.
Measure: Geometric Mean (Inter-Quartile Range); unit: months
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 31 | 1 | 17
months | 1.84 [1.77 to 1.87] | 1.74 [1.74 to 1.74] | 1.87 [1.81 to 5.16]

6. Secondary Outcome: Enrolled Population: Clinical Benefit Rate (CBR): Percentage of Participants Who Achieve CR, PR, or Stable Disease (SD) With a Duration of At Least 16 or More Weeks as Assessed by IRC
Description: CBR based on the percentage of participants with best overall response of CR, PR, or stable disease (SD) lasting 16 or more weeks following initiation of selpercatinib as assessed by IRC. CR is defined as disappearance of all target lesions. Any pathologic nodes (whether target or non-target lesions) must have a reduction in short axis diameter (SAD) to less than 10 mm. PR is defined as at least a 30% decrease in the sum of the diameters (SOD) (LD for non-nodal lesions) and SAD for nodal lesions) of target lesions, taking as reference the baseline sum LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline through Disease Progression or Death Due to Any Cause (Up to 12 Months)
Population: All eligible participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 47 | 1 | 29
percentage of participants | 76.6 [62.0 to 87.7] | 100.0 [2.5 to 100.0] | 65.5 [45.7 to 82.1]

7. Secondary Outcome: Enrolled Population: Progression Free Survival (PFS) as Assessed by IRC
Description: PFS is defined as the number of months elapsed between the date of the first dose and the earliest date of documented disease progression or death (whatever the cause). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest sum on study) for target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5.0 mm. Progressive disease for non-target lesion is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to Progressive Disease or Death from Any Cause (Up to 12 Months)
Population: All eligible participants. Number of participants censored: All NSCLC = 40; All TC = 1, and All MTC = 28
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 47 | 1 | 29
months | NA [NA to NA] — Median and CI not available due to censoring. | NA [NA to NA] — Median and CI not available due to censoring. | NA [NA to NA] — Median and CI not available due to censoring.

8. Secondary Outcome: Enrolled Population: Overall Survival (OS)
Description: OS is defined as the number of months elapsed between the date of the first dose and the date of death (whatever the cause). Participants who are alive or lost to follow-up as of the data cutoff date will be right-censored.
Time Frame: Baseline to Date of Death from Any Cause (Up to 12 Months)
Population: All eligible participants. Number of participants censored: All NSCLC = 42, All TC = 1, and All MTC = 28.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All NSCLC | All TC | All MTC
Number analyzed (Participants) | 47 | 1 | 29
months | NA [NA to NA] — Median and CI not available due to censoring. | NA [NA to NA] — Median and CI not available due to censoring. | NA [NA to NA] — Median and CI not available due to censoring.

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Selpercatinib
Description: Serial blood samples for intensive PK monitoring will be collected for 12 participants.
Time Frame: PK: Cycle 1 Day 1: Predose, 1 h, 2, h, 4 h, 8 h, 12 h postdose PK: Cycle 1 Day 8: Predose, 1 h, 2, h, 4 h, 8 h postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable intensive PK data per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Arm/Group | Selpercatinib
Number analyzed (Participants) | 12
nanogram * hour per milliliter (ng*h/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 11700 (56.8)
  Cycle 1 Day 8 | 37900 (54)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 Months
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Selpercatinib: 160 mg Selpercatinib administered orally twice daily (BID).
Arm/Group | Selpercatinib
All-Cause Mortality (participants affected / at risk) | 3/77
Serious Adverse Events (participants affected / at risk) | 17/77
Other Adverse Events (participants affected / at risk) | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Selpercatinib (N=77)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3)
Jaundice (Hepatobiliary disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/44 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1/44 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selpercatinib (N=77)
Anaemia (Blood and lymphatic system disorders) | 13 (14)
Leukopenia (Blood and lymphatic system disorders) | 5 (9)
Neutropenia (Blood and lymphatic system disorders) | 5 (8)
Sinus bradycardia (Cardiac disorders) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 6 (7)
Hypothyroidism (Endocrine disorders) | 8 (11)
Thyroid disorder (Endocrine disorders) | 8 (12)
Ascites (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 25 (136)
Dry mouth (Gastrointestinal disorders) | 22 (23)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 5 (8)
Chest pain (General disorders) | 6 (7)
Face oedema (General disorders) | 5 (5)
Fatigue (General disorders) | 8 (9)
Oedema peripheral (General disorders) | 6 (8)
Pyrexia (General disorders) | 17 (22)
Swelling face (General disorders) | 5 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (9)
Hypersensitivity (Immune system disorders) | 9 (9)
Adenosine deaminase increased (Investigations) | 4 (4)
Alanine aminotransferase increased (Investigations) | 50 (73)
Aspartate aminotransferase increased (Investigations) | 47 (83)
Bilirubin conjugated increased (Investigations) | 20 (34)
Blood alkaline phosphatase increased (Investigations) | 21 (32)
Blood bilirubin increased (Investigations) | 30 (69)
Blood bilirubin unconjugated increased (Investigations) | 6 (8)
Blood creatinine increased (Investigations) | 18 (30)
Blood lactate dehydrogenase increased (Investigations) | 18 (33)
Blood thyroid stimulating hormone increased (Investigations) | 9 (13)
Blood urea increased (Investigations) | 5 (7)
Electrocardiogram qt prolonged (Investigations) | 19 (34)
Electrocardiogram t wave abnormal (Investigations) | 10 (12)
Electrocardiogram t wave amplitude decreased (Investigations) | 5 (6)
Gamma-glutamyltransferase increased (Investigations) | 17 (23)
Globulins decreased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 9 (13)
Neutrophil count decreased (Investigations) | 20 (41)
Platelet count decreased (Investigations) | 29 (47)
Protein total decreased (Investigations) | 12 (27)
Thyroxine increased (Investigations) | 5 (6)
Total bile acids increased (Investigations) | 10 (17)
Tri-iodothyronine decreased (Investigations) | 5 (6)
Urine bilirubin increased (Investigations) | 5 (7)
Weight decreased (Investigations) | 7 (9)
Weight increased (Investigations) | 18 (25)
White blood cell count decreased (Investigations) | 25 (39)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (17)
Hyperphosphataemia (Metabolism and nutrition disorders) | 11 (21)
Hyperuricaemia (Metabolism and nutrition disorders) | 19 (36)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26 (40)
Hypocalcaemia (Metabolism and nutrition disorders) | 14 (19)
Hypochloraemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (6)
Proteinuria (Renal and urinary disorders) | 15 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 12 (13)
Hypertension (Vascular disorders) | 27 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04280081/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT04280081/SAP_001.pdf